CLINICAL TRIAL: NCT05398497
Title: Evaluation of Cryoablation in the Local Treatment of Early Breast Cancer
Brief Title: FreezIng bReaST Cancer in Brazil: a Before-after Study
Acronym: FIRST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIRST
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: cryoablation, cryotherapy, breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early stage breast cancer up to 2.5 cm (Experimental): Patients treated with Cryocare SL followed by traditional surgery, radiotherapy and adjuvant systemic therapy.
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — Cryoablation will be performed under ultrasound guidance.

SUMMARY:
Image-guided tumor ablation is a non-surgical, minimally invasive therapy available for local therapy of some carcinomas as an alternative to surgical treatment. This study assesses whether cryoablation can be used as an alternative to surgery in cases of early invasive breast carcinoma.

DETAILED DESCRIPTION:
Purpose: To evaluate the effectiveness of cryoablation in the local treatment of breast cancer, through the absence of neoplastic cells (invasive or in situ).

Outline

1. Core biopsy
2. Mammogram
3. Magnetic resonance imaging
4. Ultrasound
5. Tumor Cryoablation
6. Mammogram (post-cryoablation)
7. Magnetic resonance imaging (post-cryoablation)
8. Ultrasound (post-cryoablation)
9. Surgery
10. Evaluation of outcomes

ELIGIBILITY:
Inclusion Criteria:

* Unifocal primary invasive breast carcinoma
* Pathological report should be complete (with the result of ER, PR , HER2, KI67 and FISH report of ERBB2 gene if necessary)
* Maximum tumor size ≤2.5 cm in its greatest diameter
* Ultrasound visible lesion

Exclusion Criteria:

* Multifocal or multicentric invasive breast carcinoma
* Ductal carcinoma in-situ
* Breast cancer with skin involvement
* Clinically positive axilla (N1, N2 or N3)
* Distance from lesion and skin less than 5 mm
* Prior neoadjuvant systemic therapy for breast cancer
* Distant metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Tumor ablation | 1 month
  Successful tumor ablation will be defined as absence of residual viable invasive or in situ carcinoma in the surgical specimen.

SECONDARY OUTCOMES:
Negative predictive value of magnetic resonance imaging (MRI) | 14 days and 28 days
  Magnetic resonance imaging will be conducted between 14 to 28 days after cryoablation. Negative predictive value of MRI will be calculated according to the pathological report after the traditional surgery. Negative predictive value = number of the patients who is pathologically negative divided by the number of patients who is MRI negative.
Accuracy of conventional imaging methods (mammography and ultrasound) | 14 days and 28 days
  Mammography and ultrasound will be conducted between 14 to 28 days after cryoablation. Accuracy of conventional imaging methods will be calculated according to the pathological report after the traditional surgery.
Measurement of the ice ball by ultrasound | 14 days and 28 days
  To compare the baseline tumor size, ultrasound measurement of the ice ball, and the pathological result.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre B Cavalcanti, PhD, Study Director — Hospital do Coracao; Bruna MP Vianna, Principal Investigator — Hospital do Coracao; Vanessa M Sanvido, PhD, Principal Investigator — Hospital do Coracao; Afonso CP Nazário, Professor, Principal Investigator — Hospital do Coracao
Locations (1):
- Hcor, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to share IPD in the article publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code